CLINICAL TRIAL: NCT03738215
Title: A Double-Blind, Placebo-Controlled Study of Cariprazine as an Adjunct to Antidepressants in the Treatment of Patients With Major Depressive Disorder Who Have Had an Inadequate Response to Antidepressants Alone
Brief Title: Efficacy, Safety and Tolerability of Cariprazine as an Adjunctive Treatment to Antidepressant Therapy (ADT) in Patients With Major Depressive Disorder (MDD) Who Have Had an Inadequate Response to Antidepressants Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3111-301-001; 2018-002782-19 (EudraCT Number)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cariprazine 1.5 mg/Day + ADT (Experimental): During the double blind treatment period (6 weeks), participants will take 1 capsule of cariprazine 1.5mg, orally, per day in addition to their ongoing ADT (Same antidepressant and dose of ADT they were on at the Visit 2 baseline).
  Interventions: Drug: Cariprazine
- Cariprazine 3 mg/Day + ADT (Experimental): During the double blind treatment period (6 weeks), participants will take 1 capsule of cariprazine 1.5mg, orally, per day for two weeks in addition to their ongoing ADT (Same antidepressant and dose of ADT they were on at the Visit 2 baseline). They will then titrate to Cariprazine 3 mg, orally per day, in addition to their ADT starting at Visit 4 (Week 2).
  Interventions: Drug: Cariprazine
- Placebo + ADT (Placebo Comparator): During the double blind treatment period (6 weeks), participants will take 1 capsule of placebo, orally, per day in addition to their ongoing ADT (Same antidepressant and dose of ADT they were on at the Visit 2 baseline).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Cariprazine supplied in capsules
  Arms: Cariprazine 1.5 mg/Day + ADT; Cariprazine 3 mg/Day + ADT
Drug: Placebo — Placebo supplied in capsules
  Arms: Placebo + ADT

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and tolerability of cariprazine as an adjunctive treatment to antidepressant therapy (ADT) in patients with MDD who have had an inadequate response to antidepressants alone.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained.
* Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable (eg, Written Authorization for Use and Release of Health and Research Study Information [US sites] and written Data Protection consent [EU sites]).
* Patient must be an outpatient at the time of Visit 1 (Screening).
* Patient meets the DSM-5 criteria for MDD based on SCID-5, with a current major depressive episode of at least 8 weeks and not exceeding 24 months in duration at Visit 1/Screening. A diagnosis of MDD with psychotic features will be acceptable.
* Diagnosis of MDD confirmed through a formal adjudication process.
* Patient demonstrates ability to follow study instructions and likely to complete all required visits.
* Patient must have an inadequate response, as measured by the modified ATRQ, to 1 to 3 antidepressants administered during the current episode at an adequate dose (as per package insert) and for at least 6 weeks duration, with at least one dose escalation during the current depressive episode.
* Only one antidepressant (of sufficient dose per package insert and taken for at least 6 weeks) will be allowed at randomization and patients must agree to continue taking the same ADT dosing regimen through completion of Visit 6/ET. Patients who are taking more than one antidepressant at Screening, regardless of the indication, will need to discontinue all other antidepressants prior to Visit 2 (Baseline).
* Male and female patients must agree to use a medically acceptable and highly effective method of birth control during the course of the entire study.
* Women of childbearing potential (only) must have a negative serum β-human chorionic gonadotropin pregnancy test prior to Visit 2.

Exclusion Criteria:

* Diagnosis of any current psychiatric diagnosis other than MDD (including those with current intellectual development disability) with the exception of specific phobias.
* Patient has a history of intolerance or hypersensitivity to cariprazine or other drugs of the same class or to rescue medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbvie INC., Study Director — AbbVie
Locations (125):
- United States (65):
  - Alea Research /ID# 234789, Phoenix, Arizona
  - Atria Clinical Research /ID# 237988, Little Rock, Arkansas
  - Woodland Research Northwest, LLC /ID# 236641, Rogers, Arkansas
  - California Pharmaceutical Research Institute /ID# 236732, Anaheim, California
  - Advanced Research Center /ID# 237957, Anaheim, California
  - Axiom Research /ID# 236268, Colton, California
  - ATP Clinical Research, Inc /ID# 236619, Costa Mesa, California
  - ProScience Research Group /ID# 236442, Culver City, California
  - Collaborative Neuroscience Research - Orange County /ID# 237639, Garden Grove, California
  - Irvine Clinical Research /ID# 237409, Irvine, California
  - Omega Clinical Trials LLC /ID# 238168, La Habra, California
  - Synergy San Diego /ID# 236654, Lemon Grove, California
  - Anderson Clinical Research /ID# 236627, Redlands, California
  - Sharp Mesa Vista Hospital /ID# 235797, San Diego, California
  - Viking Clinical Research /ID# 236614, Temecula, California
  - Olympian Clinical Research /ID# 237417, Clearwater, Florida
  - MD Clinical, Hallandale, Florida
  - Reliable Clinical Research /ID# 234786, Hialeah, Florida
  - CNS Healthcare - Jacksonville /ID# 238241, Jacksonville, Florida
  - Space Coast Neuropsychiatric Research Institute /ID# 235765, Palm Bay, Florida
  - University of South Florida /ID# 234386, Tampa, Florida
  - Institute for Advanced Medical Research /ID# 236672, Alpharetta, Georgia
  - iResearch Atlanta, LLC /ID# 237389, Decatur, Georgia
  - Psych Atlanta /ID# 235835, Marietta, Georgia
  - Capstone Clinical Research /ID# 236546, Libertyville, Illinois
  - Pillar Clinical Research /ID# 235702, Lincolnwood, Illinois
  - NeuroPsychiatric Research Practice & Associate LTD /ID# 234636, Winfield, Illinois
  - Lake Charles Clinical Trials /ID# 237723, Lake Charles, Louisiana
  - J. Gary Booker MD APMC /ID# 234514, Shreveport, Louisiana
  - Pharmasite Research, Inc. /ID# 237395, Baltimore, Maryland
  - CBH Health LLC /ID# 234536, Gaithersburg, Maryland
  - Michigan Clinical Research Institute /ID# 234792, Ann Arbor, Michigan
  - NeuroBehavioral Medicine Group /ID# 236671, Bloomfield Hills, Michigan
  - Precise Research Centers /ID# 236598, Flowood, Mississippi
  - Millennium Psychiatric Associates LLC /ID# 235989, St Louis, Missouri
  - Alivation Research /ID# 236583, Lincoln, Nebraska
  - Altea Research Institute /ID# 236726, Las Vegas, Nevada
  - Hassman Research Institute /ID# 237501, Berlin, New Jersey
  - Integrative Clinical Trials /ID# 236656, Brooklyn, New York
  - Manhattan Behavioral Medicine PLLC /ID# 236314, New York, New York
  - Finger Lakes Clinical Research /ID# 236578, Rochester, New York
  - New Hope Clinical Research Inc. /ID# 234557, Charlotte, North Carolina
  - Richard Weisler MD, PA & Assoc /ID# 237424, Raleigh, North Carolina
  - Quest Therapeutics of Avon Lake /ID# 236282, Avon Lake, Ohio
  - CTI Clinical Trial and Consulting /ID# 236271, Cincinnati, Ohio
  - The Ohio State University Department of Psychiatry /ID# 234583, Columbus, Ohio
  - CincyScience /ID# 236391, West Chester, Ohio
  - IPS Research Company /ID# 237671, Oklahoma City, Oklahoma
  - Sooner Clinical Research /ID# 236346, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc. - Portland /ID# 236649, Portland, Oregon
  - Lehigh Center for Clinical Research /ID# 236702, Allentown, Pennsylvania
  - Coastal Carolina Research Center /ID# 235909, North Charleston, South Carolina
  - Psychiatric Consultants PC /ID# 235839, Franklin, Tennessee
  - Clinical Neuroscience Solutions - Memphis /ID# 237476, Memphis, Tennessee
  - Austin Clinical Trial Partners /ID# 236551, Austin, Texas
  - BioBehavioral Research of Austin /ID# 236477, Austin, Texas
  - Houston Clinical Trials /ID# 234442, Bellaire, Texas
  - FutureSearch Trials of Dallas, LP /ID# 236275, Dallas, Texas
  - Earle Research /ID# 236661, Friendswood, Texas
  - Red Oak Psychiatry Associates /ID# 236600, Houston, Texas
  - AIM Trials /ID# 236369, Plano, Texas
  - Pillar Clinical Research LLC /ID# 234465, Richardson, Texas
  - Neuropsychiatric Associates LLC/DBA Woodstock Research Center /ID# 236087, Woodstock, Vermont
  - Northwest Clinical Research Center /ID# 237584, Bellevue, Washington
  - Core Clinical Research /ID# 236405, Everett, Washington
- Bulgaria (15):
  - UMHAT Alexandrovska EAD /ID# 237834, Sofiya, Sofia
  - State Psychiatry Hospital-Kardzhali; Third Male Department /ID# 234625, Kardzhali
  - MHAT Dr. Hristo Stambolski EOOD; Hospital Pharmacy /ID# 234773, Kazanlak
  - UMHAT Dr Georgi Stranski EAD /ID# 237828, Pleven
  - Medical Center Mentalcare OOD /ID# 234934, Plovdiv
  - Clinic of Psychiatry /ID# 235878, Plovdiv
  - Mental health Centre-Ruse EOOD /ID# 234775, Rousse
  - Medical Center Sveti Naum EOOD /ID# 236069, Sofia
  - Medical Center Hera EOOD /ID# 235859, Sofia
  - Medical complex Doverie /ID# 238307, Sofia
  - Medical Centre - VAS OOD /ID# 235719, Targovishte
  - Diagnostic consultative center Mladost M /ID# 236253, Varna
  - Diagnostic consultative center Mladost M /ID# 236254, Varna
  - Mental Health Center - Veliko Tarnovo EOOD Veliko Tarnovo /ID# 236078, Veliko Tarnovo
  - Mental Health Center - Vratsa EOOD Hospital Pharmacy /ID# 235960, Vratsa
- Estonia (4):
  - Tartu University Hospital /ID# 237079, Tartu, Tartu
  - West Tallinn Central Hospital /ID# 237078, Tallinn
  - Marienthali Kliinik /ID# 235677, Tallinn
  - OU Jaanson and Laane /ID# 234985, Tartu
- Germany (8):
  - Universitaetsklinikum Frankfurt /ID# 237292, Frankfurt am Main, Hesse
  - Private Practice - Dr. Thomsen /ID# 235713, Berlin
  - Emovis GmbH /ID# 235010, Berlin
  - MVZ LIO Berlin /ID# 235711, Berlin
  - BAG Prof. Dr. Kunte / Dr. sc. med. A. Schulze /ID# 235970, Berlin
  - Arztpraxis Dr Kirsten Hahn /ID# 235958, Berlin
  - Klinikum Chemnitz gGmbH /ID# 237758, Chemnitz
  - Studienzentrum Nord-West /ID# 236357, Westerstede
- Hungary (10):
  - PsychoTech Kft. /ID# 235008, Pécs, Baranya
  - Bacs-Kiskun Megyei Oktatokorhaz Szent-Kereszt Korhaz /ID# 235974, Kalocsa, Bács-Kiskun county
  - Bugat Pal Korhaz /ID# 238145, Gyöngyös, Heves County
  - Szent Borbala Korhaz /ID# 238293, Tatabánya, Komárom-Esztergom
  - Obudai Egeszsegugyi Centrum Kft. /ID# 237495, Budapest, Pest County
  - Clinexpert Kft /ID# 237266, Budapest
  - Jozsefvarosi Szent Kozma Egeszsegugyi Kozpont /ID# 235095, Budapest
  - Semmelweis Egyetem /ID# 237096, Budapest
  - Nyiro Gyula Orszagos Pszichiatriai és Addiktologiai Intezet /ID# 235912, Budapest
  - Varoskapu Rendelo - Processus Kft. /ID# 235170, Budapest
- Ukraine (16):
  - Cherkasy regional psychiatric hospital of the CRC /ID# 234513, Smila, Cherkasy Oblast
  - Geikivka multidisciplinary hospital for psychiatric care /ID# 234498, Kryvbas Village, Dnipropetrovsk Oblast
  - KNP Prykarpatskyi Regional Clinical Centre of Mental Health /ID# 234999, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - SI Institution Neurology Psychiatry and Narcology NAMS of Ukraine /ID# 236336, Kharkiv, Kharkivs’ka Oblast’
  - SI Institution Neurology Psychiatry and Narcology NAMS of Ukraine /ID# 236338, Kharkiv, Kharkivs’ka Oblast’
  - SI Institution Neurology Psychiatry and Narcology NAMS of Ukraine /ID# 236340, Kharkiv, Kharkivs’ka Oblast’
  - Kherson Regional Psychiatric Institution for Psychiatric Care /ID# 234509, Stepanivka Village, Kherson Oblast
  - Odesa regional psychiatric hospital 2 of the ORC /ID# 234505, Oleksandrivka Village, Odesa Oblast
  - KNP Zakarpatskyi Regional MC of Mental Health and Medicine of Dependencies /ID# 234499, Uzhhorod, Zakarpattia Oblast
  - KNP Kyiv City Psychoneurological Hospital /ID# 235093, Kyiv
  - Kyiv Railway Clinical Hosp No.2 /ID# 237405, Kyiv
  - CNE of LOR Lviv Regional Clinical Psychiatric Hospital /ID# 236270, Lviv
  - MNCE Odesa Regional Medical Center for Mental Health /ID# 235723, Odesa
  - Ternopil University Hospital /ID# 236819, Ternopil
  - Vinnytsia Regional Psycho-Neurological Hospital /ID# 235178, Vinnytsia
  - Vinnytsia Regional Psycho-Neurological Hospital /ID# 235179, Vinnytsia
- United Kingdom (7):
  - Knowle House Surgery /ID# 235025, Plymouth, Devon
  - St. Peter's Hospital Surrey and Borders Partnership NHS FT /ID# 235725, Chertsey, Surrey
  - MAC Clinical Research /ID# 235938, Blackpool
  - MAC Clinical Research /ID# 235941, Blackpool
  - MAC Clinical Research /ID# 235945, Blackpool
  - MAC Clinical Research /ID# 239078, Blackpool
  - MAC Clinical Research-Manchester /ID# 235940, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Sachs GS, Yeung PP, Rekeda L, Khan A, Adams JL, Fava M. Adjunctive Cariprazine for the Treatment of Patients With Major Depressive Disorder: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study. Am J Psychiatry. 2023 Mar 1;180(3):241-251. doi: 10.1176/appi.ajp.20220504. Epub 2023 Feb 15. PMID 36789515

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 759 participants were randomized to double-blind treatment, 757 participants received at least 1 dose of double-blind investigational product (safety population), and 751 treated participants had at least 1 postbaseline assessment of MADRS total score (modified intent-to-treat [mITT] population ). At the end of treatment in the Double-blind Period, participants continued on their background antidepressant therapy (ADT) and entered the Safety Follow-up Period.
Period: Double-blind Treatment Period (6 Weeks)
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Started | 253 | 252 | 252
Completed | 229 | 231 | 219
Not Completed | 24 | 21 | 33
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 2 | 0
Not completed — Adverse Event | 6 | 3 | 18
Not completed — Withdrawal by Subject | 13 | 11 | 9
Not completed — Non-Compliance with Study Drug | 0 | 1 | 1
Not completed — Lost to Follow-up | 3 | 3 | 5
Period: Safety Follow Up Period (4 Weeks)
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Started | 240 | 239 | 238
Completed | 237 | 234 | 230
Not Completed | 3 | 5 | 8
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Reason Not Specified | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Lost to Follow-up | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants in the randomized population who took ≥ 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT | Total
Number analyzed (Participants) | 253 | 252 | 252 | 757
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.89) | 43.3 (13.59) | 44.8 (13.33) | 44.8 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 191 | 180 | 555
  Male | 69 | 61 | 72 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 24 | 19 | 68
  Not Hispanic or Latino | 228 | 228 | 233 | 689
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 5 | 4 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 0 | 4
  Black or African American | 43 | 37 | 30 | 110
  White | 203 | 205 | 215 | 623
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 152 | 153 | 153 | 458
  Bulgaria | 35 | 34 | 34 | 103
  Estonia | 10 | 10 | 9 | 29
  Germany | 13 | 12 | 12 | 37
  Hungary | 7 | 7 | 7 | 21
  Ukraine | 33 | 33 | 34 | 100
  United Kingdom | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Total Score Change From Baseline to Week 6 in the MADRS (Montgomery-Åsberg Depression Rating Scale)
Description: The MADRS is a 10-item, clinician-rated scale that evaluates the patient's depressive symptomatology during the past week. Patients are rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item is scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity. mITT Population included all randomized participants who had ≥1 postbaseline assessment of the MADRS total score. Number of subjects analyzed are the number of participants with data available for analyses.
Time Frame: Baseline and Week 6
Population: mITT population includes all randomized participants who had ≥ 1 postbaseline assessment of the MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Number analyzed (Participants) | 231 | 231 | 223
score on a scale | -11.5 (0.70) | -14.1 (0.70) | -13.1 (0.70)
Statistical Analysis 1: Comparison: Placebo + ADT vs Cariprazine 1.5 mg/Day + ADT; Test type: Superiority; p = 0.0050, MMRM — Adjusted P-Value (based on truncated Hochberg with parameter=0.9); MMRM = mixed-effects model for repeated measures; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-4.17 to -0.89]
Statistical Analysis 2: Comparison: Placebo + ADT vs Cariprazine 3 mg/Day + ADT; Test type: Superiority; p = 0.0727, MMRM — Adjusted P-Value (based on truncated Hochberg with parameter=0.9); MMRM = mixed-effects model for repeated measures; Least Squares Mean Difference = -1.5, 95% CI 2-sided [-3.16 to 0.12]

2. Secondary Outcome: Change From Baseline to Week 6 in the Clinical Global Impressions-Severity (CGI-S) Score
Description: The CGI-S is a clinician-rated scale used to rate the severity of the participant's current state of mental illness compared with MDD population. The participant was rated on a scale from 1 to 7, where 1=normal, not at all ill and 7=among the most extremely ill participants. Higher scores indicate worsening of mental illness. A negative change from Baseline indicates improvement. MMRM was used for analyses. mITT Population included all randomized participants who had ≥1 postbaseline assessment of the MADRS total score. Number of subjects analyzed are the number of participants with data available for analyses.
Time Frame: Baseline and Week 6
Population: mITT population includes all randomized participants who had ≥ 1 postbaseline assessment of the MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Number analyzed (Participants) | 231 | 231 | 223
score on a scale | -1.1 (0.09) | -1.4 (0.09) | -1.3 (0.09)
Statistical Analysis 1: Comparison: Placebo + ADT vs Cariprazine 1.5 mg/Day + ADT; Test type: Superiority; p = 0.0727, MMRM — Adjusted P-Value (based on Hochberg procedure); MMRM = mixed-effects model for repeated measures; Lease Squares Mean Difference = -0.3, 95% CI 2-sided [-0.49 to -0.07]
Statistical Analysis 2: Comparison: Placebo + ADT vs Cariprazine 3 mg/Day + ADT; Test type: Superiority; p = 0.0944, MMRM — Adjusted P-Value (based on Hochberg procedure); MMRM = mixed-effects model for repeated measures; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.39 to 0.03]

ADVERSE EVENTS:
Time Frame: First Dose of study drug until 30 days after the last dose of study drug (up to 12 weeks)
Description: Safety Population included all participants in the randomized population who took ≥ 1 dose of double-blind investigational product.
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/252 | 0/252
Serious Adverse Events (participants affected / at risk) | 2/253 | 3/252 | 3/252
Other Adverse Events (participants affected / at risk) | 39/253 | 68/252 | 62/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + ADT (N=253) | Cariprazine 1.5 mg/Day + ADT (N=252) | Cariprazine 3 mg/Day + ADT (N=252)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
SOCIAL STAY HOSPITALISATION (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + ADT (N=253) | Cariprazine 1.5 mg/Day + ADT (N=252) | Cariprazine 3 mg/Day + ADT (N=252)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 20 (21) | 16 (19)
AKATHISIA (Nervous system disorders) | 3 (3) | 13 (14) | 20 (23)
HEADACHE (Nervous system disorders) | 16 (19) | 24 (25) | 11 (23)
SOMNOLENCE (Nervous system disorders) | 7 (7) | 13 (13) | 11 (12)
INSOMNIA (Psychiatric disorders) | 11 (18) | 18 (18) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT03738215/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT03738215/SAP_001.pdf